CLINICAL TRIAL: NCT06440161
Title: Association of Intraoperative Haemodynamic Instability With Postoperative Mortality, Renal Injury, and Stroke in Type A Aortic Dissection Surgery: A Retrospective Cohort Analysis
Brief Title: Association of Intraoperative Haemodynamic and Postoperative Complications in Type A Aortic Dissection Surgery
Status: Completed | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20230918-KS-02
Record Dates: First submitted 2024-05-06; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2023-09

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Intraoperative Hypotension; Venous Congestion; Acute Kidney Disease; Type A Aortic Dissection
MeSH Terms: conditions — Acute Kidney Injury; Hyperemia | interventions — COP protocol 2; Arterial Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Primary exposures were venous congestion defined by central venous pressure (CVP) and mean arterial pressure (MAP). — After the induction of anaesthesia, a central venous or pulmonary artery catheter was positioned. Based on prior studies, thresholds for central venous pressure were set at 10, 12, 16, and 20 mm Hg. Venous congestion was quantified by time exceeding each CVP threshold and the area under the curve (AUC) surpassing each CVP threshold in mmHg × min. Assessments were limited to pre- and post-CPB periods, as the venous drainage cannulate generated negative CVP during CPB.
  An arterial catheter was installed upon room admission. Continuous arterial blood pressure monitoring commenced after exposure to atmospheric pressure and calibration to zero. The MAP was determined using the formula: 2/3 × diastolic blood pressure + 1/3 × systolic blood pressure. Data were logged by automated software every minute. Established thresholds for MAP were 55, 65, and 75 mm Hg. Hypotension was quantified as (1) time under each MAP threshold in minutes and (2) the AUC below each MAP threshold in mmHg × min.

SUMMARY:
Background To determine whether venous congestion is an important predictor of postoperative kidney injury and other adverse events after type A aortic dissection (TAAD).

Methods Authors collected data of adults who underwent surgery for TAAD between January 2016 and July 2023. Primary exposures were venous congestion defined by central venous pressure (CVP) and mean arterial pressure (MAP). The primary outcomes were acute kidney injury (AKI) and acute injury disease (AKD). The secondary outcomes encompassed death and stroke. Restricted cubic spline regression model was used to adjust for confounding factors and multiple comparisons.

DETAILED DESCRIPTION:
Type A aortic dissection (TAAD) is a catastrophic cardiac macrovascular disease with a striking in-hospital mortality rate of 22%-31%. Among the myriad of complications following TAAD surgeries, acute kidney injury (AKI) is one of the most prevalent, boasting an incidence of 40-55%. Notably, this incidence surpasses that observed in other cardiovascular procedures, such as coronary artery bypass grafting (CABG), which ranges from 10-20%, and aortic valve replacement (AVR) at 17-23%. Furthermore, the occurrence of AKI post-TAAD surgeries has been linked with escalated in-hospital, short-term, and long-term mortalities, as well as significant complications.

Preoperatively, patients with TAAD usually have poorly controlled blood pressure, long-term hypertension can cause chronic kidney damage. In some cases, involving renal artery origins, renal perfusion insufficiency may exist preoperatively. Intraoperatively, the kidneys need to undergo a complete ischemic phase of deep hypothermic circulatory arrest (DHCA), inflammatory reactions associated with cardiopulmonary bypass (CPB), and a large number of blood and fluid transfusions could potentially cause renal dysfunction. Patients are at high risk for postoperative surgical site infection following TAAD procedure, further exacerbating acute kidney injury. The myriad factors mentioned above collectively exacerbate the elevated occurrence of kidney injury following Type A Aortic Dissection (TAAD) surgeries when juxtaposed with other cardiac surgical procedures. Pathological anatomy and surgical procedure intricacies pose formidable challenges in mitigation. Consequently, the pursuit of precise intraoperative hemodynamic management objectives aimed at maximizing organ perfusion has emerged as a focal point in contemporary research endeavours. A study encompassing 5,127 patients undergoing CABG and cardiac valvular surgery underscored the role of venous congestion duration and severity as independent postoperative AKI/AKD risk determinants. However, the relationship between intraoperative hemodynamic in TAAD surgeries and ensuing AKI/AKD remains elusive. There's a paucity of comprehensive evaluations, primarily due to a dearth of long-term data from expansive TAAD cohorts. The investigators' primary objective was to discern the correlation between intraoperative hypotension and venous congestion durations and magnitudes at varied thresholds during TAAD surgeries and the subsequent risks of postoperative AKI/AKD. As a secondary objective, the investigators sought to elucidate the association between intraoperative hemodynamic and major adverse events, including stroke and mortality. The investigators hypothesize that both intraoperative hypotension and venous congestion are paramount predictors for postoperative AKI and AKD following TAAD surgeries.

ELIGIBILITY:
Inclusion Criteria:

1) Eligible patients were adults, aged 18 or older.

Exclusion Criteria:

1. Lacking preoperative serum creatinine (Scr) values
2. Insufficient hemodynamic or laboratory data
3. Exhibiting a preoperative Scr level ≥133 μmol/L
4. Patients with renal insufficiency before surgery
5. Patients on preoperative dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients underwent surgery for TAAD.
Sampling Method: Non-Probability Sample
Enrollment: 543 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
The Incidence of AKI | After the surgery，up to 7 days
  AKI diagnosis adhered to the Kidney Disease Improvement Global Prognosis Organization (KDIGO) criteria.
The Incidence of AKD | After the surgery，longer than 7 days but within 90 days
  AKD staging was determined based on the Acute Disease Quality Initiative (ADQI) Working Group consensus, using available Scr values from 8 to 90 days post-surgery.

SECONDARY OUTCOMES:
The days of stay in hospital | perioperatively
  The days of stay in hospital
The days of stay in ICU | after surgery
  The days of stay in ICU
The incidence of in-hospital mortality | after surgery
  The incidence of in-hospital mortality
The incidence of 30-day all-cause mortality | after surgery
  The incidence of 30-day all-cause mortality
The incidence of stroke | after surgery
  Stroke diagnosis adhered to National Institute of Neurological Disorders and Stroke rt PA Stroke study Group

CONTACTS AND LOCATIONS:
Overall Officials: Ya-li Ge, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No